CLINICAL TRIAL: NCT02473250
Title: Prediction of Clinical Response to SSRI Treatment in Bipolar Disorder Using Serotonin 1A Receptor PET Imaging
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Martin Lan, Clinical Psychiatrist, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: #7056
Record Dates: First submitted 2015-06-10; First posted 2015-06-16 (Estimated); Results first posted 2021-04-01 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Fluoxetine; Citalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bipolar depressed (Experimental): Bipolar depressed subjects will have neuroimaging and treatment with fluoxetine in combination with a mood stabilizer (valproate)
  Interventions: Drug: Fluoxetine; Drug: Citalopram

INTERVENTIONS:
Drug: Fluoxetine — Bipolar depressed patients will be treated with fluoxetine in combination with a mood stabilizer (valproate).
  Other Names: Prozac
Drug: Citalopram — Bipolar depressed patients will be treated with citalopram in combination with a mood stabilizer (valproate) if fluoxetine is not clinically warranted.
  Other Names: Celexa

SUMMARY:
This study is for subjects with a diagnosis of bipolar disorder who have depression at the time of recruitment. It involves brain imaging with an MRI (magnetic resonance imaging) and PET scan (positron emission tomography) and treatment with an antidepressant. The medication involves adding an SSRI (either celexa/citalopram or prozac/fluoxetine) to a mood stabilizer.

DETAILED DESCRIPTION:
Bipolar disorder is associated with alterations of chemicals in the brain, including one named serotonin. Treatment of depression in bipolar disorder can be accomplished by increasing serotonin function by medications named selective serotonin reuptake inhibitors (SSRI's). Serotonin signals in the brain occur through receptors in a way that is similar to a lock and key, where serotonin is a key and the receptor is a lock. One important receptor is the serotonin 1A (5-HT1A) receptor. This receptor has been found to be abnormal in bipolar disorder during periods of depression, as measured by a type of brain imaging called positron emission tomography (PET). The amount of brain 5-HT1A receptor measured by imaging has also been associated with how well depressed patients with major depressive disorder respond to an SSRI medication. This project will measure the 5-HT1A receptors in bipolar depressed individuals using PET with the radiotracer [11C]-CUMI-101 and will evaluate the ability of this brain imaging signal to predict how patients respond to SSRI treatment when added to a mood stabilizer.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Diagnosis of bipolar I disorder or bipolar II disorder and currently meet criteria for a major depressive episode
* Patients who were on psychiatric medication at presentation will have failed that regimen, as defined as not achieving at least partial remission after an adequate dose of medication for at least six weeks.
* Depression of sufficient severity to score at least 16 on the first 17 items of the Hamilton Depression Rating Scale
* Age range 18-60 years
* Females of child-bearing potential must be willing to use an acceptable method of birth control throughout the study.
* Subject agrees to discontinue all psychotropic other than those in the PSF and other types of drugs likely to interact with the 5-HT1A receptors.
* Subject is likely to tolerate medication cross-taper to monotherapy with a mood stabilizer (valproate, lamotrigine or lithium).

Exclusion Criteria:

* Diagnosis of any other major psychiatric disorders such as lifetime schizophrenia, schizoaffective disorder, current psychotic depression or current drug or alcohol abuse (within two months before the study) or recent drug or alcohol dependence (within six months before the study); anorexia nervosa or bulimia nervosa within the last year; IV drug use of ecstasy use more than three times. Meet criteria for a manic episode at the time of screening.
* Previous failed trial of fluoxetine and citalopram by themselves or in combination with an anti-manic agent, defined as at least six weeks of treatment at the dose of 20 mg per day or more. Failure of two trials of any SSRI or SNRI antidepressant medications.
* If the patients are discontinuing medications as part of the washout period or are starting valproate, previous failed trial of mood stabilizer that they will take alone.
* Experienced intolerable side effects of both citalopram and fluoxetine in the past. If the subject is not on medications, intolerable side effects of valproate in the past.
* History of clinical deterioration when any of the medications that the patient is taking at presentation have been discontinued in the past with the exception of any medications that will be continued during the research protocol.
* A first-degree family history of schizophrenia if the subject is less than 33 years old
* Significant active physical illness, including blood dyscrasias, lymphomas, hypersplenism, endocrinopathies, renal failure, chronic obstructive lung disease, autonomic neuropathies, peripheral vascular disease, malignancy
* Actively suicidal, as defined by expressing ideation with a plan for suicide or develops suicidal ideation that requires immediate medication or treatment intervention.
* Pregnancy, abortion or miscarriage in the two months prior to enrollment or plans to conceive during the course of study participation
* Lactating women
* ECT within the past 6 months
* Subjects who endorse a history of prior head trauma and score 1.5 standard deviations below the mean on Trail-making A & B will be excluded from study participation.
* Metal implants, pacemaker, metal prostheses, metal orthodontic appliances or shrapnel in the body
* Current, past or anticipated exposure to radiation, including:

  * Having been badged for radiation exposure in the workplace
  * Participation in nuclear medicine protocols in the last year. Subjects will be eligible, however, if the injected dose and dosimetry of the radiotracer are known and the cumulative annual exposure of the previous study and this study is lower than the annual limit for research subjects defined by the FDA (21 CFR 361.1)
* History of claustrophobia that would prevent the participation in imaging scans
* Current anticoagulant or anti-platelet treatment other than aspirin
* Obesity with weight >350 lbs or inability to fit into the MRI scanner

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Lan, MD PHD, Principal Investigator — Columbia University
Locations (1):
- New York State Psychiatric Institute/Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Lan MJ, Pantazatos SP, Ogden RT, Rubin-Falcone H, Hellerstein D, McGrath PJ, Mann JJ. Resting State MRI Amplitude of Low Frequency Fluctuations Associated With Suicidal Ideation in Bipolar Depression. J Clin Psychiatry. 2022 Mar 30;83(3):21m14054. doi: 10.4088/JCP.21m14054. PMID 35377567
- [Derived] Lan MJ, Zanderigo F, Pantazatos SP, Sublette ME, Miller J, Ogden RT, Mann JJ. Serotonin 1A Receptor Binding of [11C]CUMI-101 in Bipolar Depression Quantified Using Positron Emission Tomography: Relationship to Psychopathology and Antidepressant Response. Int J Neuropsychopharmacol. 2022 Aug 4;25(7):534-544. doi: 10.1093/ijnp/pyac001. PMID 34996114
- See also: Related Info — http://www.bipolarimaging.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Bipolar Depressed: Bipolar depressed subjects had neuroimaging and treatment with a selective serotonin reuptake inhibitor in combination with a mood stabilizer. Fluoxetine was offered first, but citalopram was offered as an alternative if fluoxetine was not clinically appropriate.
Period: Overall Study
Arm/Group | Bipolar Depressed
Started | 40
Completed | 20
Not Completed | 20
Not completed — Lost to Follow-up | 10
Not completed — Physician Decision | 5
Not completed — Did not tolerate medication washout | 3
Not completed — Antidepressant effect of divalproex | 2

BASELINE CHARACTERISTICS:
Arm/Group | Bipolar Depressed
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 23
  More than one race | 6
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale
Description: Depression severity. Minimum=0, Maximum=60. Higher numbers correspond to greater depression severity. The percent change between week 0 and the last observation was calculated.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Percent change in MADRS from baseline
Arm/Group | Bipolar Depressed
Number analyzed (Participants) | 20
Percent change in MADRS from baseline | -39.24 (10.38)

2. Secondary Outcome: Hamilton Anxiety Rating Scale
Description: Anxiety severity. Minimum=0, Maximum=56. The larger the value on the scale, the more intense the anxiety. The percent difference between week 0 and the last observation was calculated.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Percent change in HAMA score
Arm/Group | Bipolar Depressed
Number analyzed (Participants) | 20
Percent change in HAMA score | -13.95 (70.38)

3. Secondary Outcome: Young Mania Rating Scale
Description: Measure of manic symptoms. Minimum=0, Maximum=60. The higher the value on the scale, the more intense the manic symptoms. The maximum value of YMRS over the six week clinical trial is reported.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Bipolar Depressed
Number analyzed (Participants) | 20
Scores on a scale | -5.75 (2.49)

4. Secondary Outcome: Clinical Global Impression-1
Description: General impression of symptoms by clinician. Minimum=1, Maximum=7. The higher value on the scale, the more symptomatic the patient is. The percent difference between week 0 and the last observation was calculated.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Percent change in CGI score
Arm/Group | Bipolar Depressed
Number analyzed (Participants) | 20
Percent change in CGI score | -27.17 (25.06)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the time that the participants were enrolled in the study. This time range varied depending on the research procedures performed. If all research procedures were performed, the participants were enrolled for 11 weeks.
Arm/Group | Bipolar Depressed
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 2/40
Other Adverse Events (participants affected / at risk) | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bipolar Depressed (N=40)
Psychiatric Hospitalization (Psychiatric disorders) | 2 (2) — Two patients required psychiatric hospitalization during the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-27): https://cdn.clinicaltrials.gov/large-docs/50/NCT02473250/Prot_SAP_001.pdf
  • Informed Consent Form (2019-10-25): https://cdn.clinicaltrials.gov/large-docs/50/NCT02473250/ICF_000.pdf